CLINICAL TRIAL: NCT05548127
Title: TACTIVE-U: An Interventional Safety and Efficacy Phase 1b/2, Open-label Umbrella Study to Investigate Tolerability, pk, and Antitumor Activity of Vepdegestrant (ARV-471/PF-07850327), an Oral Proteolysis Targeting Chimera, in Combination With Other Anticancer Treatments in Participants Aged 18 Years and Over With ER+ Advanced or Metastatic Breast Cancer, Sub-study A (ARV-471 in Combination With Abemaciclib)
Brief Title: TACTIVE-U: A Study to Learn About the Study Medicine (Vepdegestrant) When Given With Other Medicines in People With Advanced or Metastatic Breast Cancer (Sub-Study A)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4891006; 2022-502228-34-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-08-25; First posted 2022-09-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: TACTIVE-U; Umbrella study; PROTAC; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: Phase 1b will use an escalation/de-escalation approach to determine the RP2D of ARV-471 when administered in combination with abemaciclib. The decision to de-escalate the starting dose levels of ARV 471 will be using mTPI-2 decision criteria based on the number of DLT-evaluable participants and the number of DLTs in those participants during the DLT observation period (Cycle 1 [first 28 days]).
  Phase 2 will further evaluate the preliminary antitumor activity and safety of the combination RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARV-471 in combination with Abemaciclib (Experimental): ARV-471 administered orally once daily (QD) and Abemaciclib orally twice daily (BID) on 28-day cycle
  Interventions: Drug: ARV-471; Drug: Abemaciclib

INTERVENTIONS:
Drug: ARV-471 — Daily oral dosages of ARV-471 continuously, dose escalation/de-escalation in Phase 1b until the recommended phase 2 dose (RP2D) determined, cycles lasting 28 days
  Other Names: vepdegestrant, PF-07850327
Drug: Abemaciclib — Daily oral dosages of Abemaciclib continuously, cycles lasting 28 days

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called ARV-471) when given together with other medicines for the potential treatment of advanced or metastatic breast cancer.

This study is seeking participants who have breast cancer that:

* is advanced, may have spread to other organs (metastatic) and cannot be fully treated by surgery or radiation therapy
* is sensitive to hormonal therapy (it is called estrogen receptor positive); and
* is no longer responding to previous treatments This study is divided into separate sub-studies.

For Sub-Study A:

All participants will receive ARV-471 and a medicine called abemaciclib. ARV-471 will be given by mouth, at home, 1 time a day. Abemaciclib will be given by mouth, at home, 2 times a day. We will examine the experiences of people receiving the study medicines. This will help us determine if the study medicines are safe and effective.

Participants will continue to take ARV-471 and abemaciclib until their cancer is no longer responding, or side effects become too severe. They will have visits at the study clinic about every 4 weeks.

DETAILED DESCRIPTION:
C4891006 is a sub-study from the Umbrella platform, TACTIVE-U, comprising multiple sub-studies that independently evaluate ARV-471 in participants with Estrogen Receptor Positive (ER+) Advanced or Metastatic Breast Cancer (A/MBC). ARV-471 will act as the backbone therapy given in combination with other anticancer agents thought to have clinical relevance in ER+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* histological or cytological diagnosis of ER+ and HER2- advanced/metastatic breast cancer that is not amendable to surgical resection with curative intent (≥1% ER+ stained cells on the most recent tumor biopsy).
* prior anticancer therapies: at least 1 and no more than 2 lines of prior therapies for advanced/metastatic disease; 1 line of any CDK4/6 inhibitor-based regimen is required (independent of the setting eg, adjuvant or advanced/metastatic)
* at least 1 measurable lesion as defined by RECIST v1.1.
* ECOG PS ≤1.

Exclusion Criteria:

* visceral crisis at risk of life-threatening complications in the short term
* known history of drug-induced pneumonitis or other significant symptomatic deterioration of lung functions.
* newly diagnosed brain metastases, or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease. Participants with a history of CNS metastases or cord compression are eligible if they have been definitively treated, clinically stable and discontinued anti-seizure medications and corticosteroids for at least 14 days prior to enrollment in the study.
* history of any other tumor malignancies within the past 3 years, except for the following: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated in situ carcinoma of the cervix.
* inflammatory breast cancer
* impaired cardiovascular function or clinically significant cardiovascular diseases
* concurrent administration of medications, food, or herb supplements that are strong inhibitors and strong/moderate inducers of CYP3A and drugs known to predispose to Torsade de Pointes or QT interval prolongation.
* renal impairment, not adequate liver function and/or bone marrow function
* known active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: number of participants with dose limiting toxicities | 28 days
  Dose Limiting Toxicities rate for ARV-471 in combination with abemaciclib, estimated based on data from DLT-evaluable participants during the DLT observation period (Cycle 1 [28 days]).
Phase 2: percentage of participants with objective response by investigator assessment | Up to approximately 1 year
  Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. as determined by investigator assessment.

SECONDARY OUTCOMES:
Phase 1b and Phase 2: number of participants experiencing any AE, SAE, Treatment Related SAE | Up to 28 days after last dose of study treatment
  An adverse event (AE) were any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE is any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. Treatment-related AE is any untoward medical occurrence attributed to study drug in a participant who received study drug.
  AEs were graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE version 5.0) and coded using MedDRA were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe and Grade 4=life-threatening or disabling and grade 5=death.
Phase 1b and Phase 2: number of participants with lab abnormalities - Hematology and coagulation parameters | Up to 28 days after last dose of study treatment
  Blood samples were collected for the analysis of following hematology and coagulation parameters: hemoglobin [g/L], platelets, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils and basophils [10^9/L]; partial thromboplastin time prolonged, international normalized ratio increased, prothrombin time. Number of participants with hematological and coagulation abnormalities by grade as per CTCAE version 5.0 were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe and Grade 4=life-threatening or disabling and grade 5=death.
  For laboratory tests without CTCAE grade definitions, results will be categorized as normal, abnormal, or not done.
Phase 1b and Phase 2: number of participants with lab abnormalities - chemistry parameters | Up to 28 days after last dose of study treatment
  Blood samples were collected for analysis of clinical chemistry parameters. These included: alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, [international unit per liter (IU/L)] ; Lipase and amilase [IU/L] (limited to cycle1 only); Albumin, bilirubin, urea ,calcium, creatinine, glucose, magnesium, phosphate, uric acid, chloride, potassium and sodium [millimol per liter (mmol/L)]; eGFR [milliliter per minute (ml/min)]. Number of participants with blood chemistry abnormalities by grade as per CTCAE version 5.0 were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe and Grade 4=life-threatening or disabling and grade 5=death.
  For laboratory tests without CTCAE grade definitions, results will be categorized as normal, abnormal, or not done.
Phase 1b: percentage of participants with objective response by investigator assessment | Up to approximately 1 year
  Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. as determined by investigator assessment.
Phase 1b and Phase 2: duration of response by investigator assessment. | Up to approximately 3 years
  Duration of Response (DoR) is defined for participants with confirmed OR (CR or PR) as the time from the first documentation of OR to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Phase 1b and Phase2: Percentage of participants with Clinical Benefit Response by investigator assessment. | Up to approximately 1 year
  Clinical Benefit Response (CBR) is defined as the proportion of participants with Best Overall Response of confirmed CR or PR at any time, or Stable Disease (SD) ≥24 weeks
Phase 1b and Phase 2: Progression Free Survival by investigator assessment. | Up to approximately 3 years
  Progression Free Survival (PFS) is defined as the time from the date of first dose of study interventions to the date of first documentation of PD or death due to any cause, whichever occurs first.
Phase 2: Overall Survival | Through study completion, up to approximately 3 year
  Overall Survival (OS) is defined as the time from the date of first dose of study interventions to the date of death due to any cause
Phase 2:ctDNA plasma quantitative changes from pre-treatment | Day 1, 29 and 57 and End of Treatment (an average of 1 year)
  To assess changes from baseline levels in plasma circulating DNA (ctDNA) with treatment and to evaluate potential predictability of their associations with clinical outcome
Phase 1b: Area Under the Curve from Time Zero to end of dosing interval Evaluation of abemaciclib with or without ARV-471 | Phase 1b: pre-dose Day -1, 1, 15, 29, 43, 57, 113, 169; 1, 2, 4, 6, 8 hours post dose on Day -1 and 15; post dose Day 29 and 43
  Exposure (AUCtau) of abemaciclib with and without co-administration of ARV-471
Phase 1b: Maximum Observed Plasma Concentration (Cmax) of abemaciclib with or without ARV-471 | Phase 1b: pre-dose Day -1, 1, 15, 29, 43, 57, 113, 169; 1, 2, 4, 6, 8 hours post dose on Day -1 and 15; post dose Day 29 and 43
  Concentration (Cmax) of abemaciclib with and without co-administration of ARV-471
Phase 1b and Phase 2: Maximum Observed Plasma Concentration (Cmax) of ARV-471 | Phase 1b: pre-dose Day 1, 15, 29, 43, 57, 113, 169; 1, 2, 4, 6, 8 hours post dose on Day 15; post dose Day 29 and 43. Phase 2: pre and post dose Day 15, 29 and 43; pre - dose Day 57, 113 and 169
  Plasma concentration of ARV-471
Phase 1b and Phase 2: Maximum Observed Plasma Concentration (Cmax) of abemaciclib | Phase 1b: pre-dose Day -1, 1, 15, 29, 43, 57, 113, 169; 1, 2, 4, 6, 8 hours post dose on Day -1 and 15; post dose Day 29, 43 and 57 Phase 2: pre and post dose Day 15, 29 and 43; pre - dose Day 57, 113 and 169
  Plasma concentration of abemaciclib

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (24):
  - Stanford Women's Cancer Center, Palo Alto, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Moffitt Cancer Center - International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Richard M. Shulze Family Foundation Outpatient Center, Tampa, Florida
  - Moffitt McKinley Hospital, Tampa, Florida
  - Memorial Hospital, Shiloh, Illinois
  - Siteman Cancer Center - Shiloh, Shiloh, Illinois
  - Siteman Cancer Center - WUPI, Shiloh, Illinois
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - U.T. MD Anderson Cancer Center, Investigational Pharmacy Services - Unit 376, Houston, Texas
  - U.T. MD Anderson Cancer Center, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties, PLLC, Bonney Lake, Washington
  - Northwest Medical Specialties, PLLC, Federal Way, Washington
  - Northwest Medical Specialties, PLLC, Gig Harbor, Washington
  - Northwest Medical Specialties, PLLC, Puyallup, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Canada (5):
  - BC Cancer Vancouver, Vancouver, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Rome, Lazio
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Universitari Dexeus, Barcelona, Catalunya [cataluña]
  - Clinica Universidad de Navarra, Madrid, Madrid, Comunidad de
  - Clínica Universidad de Navarra, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891006